CLINICAL TRIAL: NCT05093283
Title: The Effect of Virtual Reality Glasses on Fetal Movement, Fetal Heart Rate, Maternal Satisfaction and Anxiety Level
Brief Title: The Effect of Virtual Reality Glasses on Fetal Movement
Acronym: Virtual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mine Gokduman Keles (Other Government)
Responsible Party: Sponsor-Investigator, Mine Gokduman Keles, professional, Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate
Organization: Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TurkishMoHKahramanmarasPH
Record Dates: First submitted 2021-09-14; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Virtual Reality
Keywords: Virtual Reality; Fetal Movement; Fetal Heart Rate; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workgroup (Experimental): The probes will be fixed by giving the left lateral position for NST to the pregnant women in the intervention group by the researcher. After providing internet connection with a smart phone for the image, by clicking on youtube.com link, Relaxation (https://www.youtube.com/watch?v=H1iboKia3AQ) nature video watching virtual reality glasses will be provided. The name and surname of the pregnant woman will be written on the NST trace and the trace will be photographed. After the NST process is completed, the NST traces will be evaluated by the researchers.
  Interventions: Device: Virtual Reality Glasses
- Control (No Intervention): Unlike the study group, only video monitoring will not be applied to the pregnant women included in the control group. Other applications will be done in the same way.

INTERVENTIONS:
Device: Virtual Reality Glasses — Virtual Reality Glasses
  Arms: Workgroup

SUMMARY:
When the literature is examined, it is seen that virtual reality glasses are used during medical procedures, have an anxiety-lowering effect and have a reducing effect on the perception of fatigue (20, 7, 10, 11). On the other hand, no study has been found in the literature on the application of virtual glasses to pregnant women who underwent NST. However, in line with the results of the study on virtual glasses, it is thought that the application of virtual glasses will also have a positive effect on the Reactive (Negative) Non-Stress Test result by reducing the anxiety level of pregnant women and increasing fetal movement and fetal cup speed in pregnant women with NST.

This study was planned to examine the effects of virtual reality glasses, one of the cognitive behavioral techniques, on fetal movement, fetal heart rate, maternal satisfaction and anxiety level.

DETAILED DESCRIPTION:
One of the parameters used in the evaluation of fetal health during pregnancy is the Non-Stress Test (NST). When a healthy fetus moves, the oxygen requirement increases, the fetus increases the cardiac output to meet this requirement, and this is reflected in the trace as acceleration. Increased fetal heart rate during fetal movements; Adequate oxygenation, healthy transmission between the fetal central nervous system and the heart, and the ability of the fetus to respond to stimuli indicate fetal well-being (4, 23). This physiological response of the fetus is evaluated with the Non-Stress Test. The best result of this test is between 30-32 days of pregnancy when the fetal central nervous system development is completed. It is applied starting from these weeks in order to evaluate fetal health in routine pregnancy follow-ups (4). The results of the Non-Stress test are evaluated under two headings: Reactive (negative) and non-reactive (positive) NST. 1) Reactive (Negative) Non-Stress Test: At least two fetal movements within 20 minutes, fetal heart rate (FKA) being more than 15 beats (increase) than basal fetal heart rate in parallel with the movements, and accelerations lasting more than 15 seconds (fetal heart rate increases). 2) Non-reactive (Positive) Non-Stress Test: It is the situation in which there are accelerations (fetal heart rate increases) that are less than 15 beats and last less than 15 seconds despite the absence of fetal movements or fetal movements (4). The expected result in a healthy fetus is the Reactive (Negative) Non-Stress Test result. In the study of one it was found that 95% of the pregnant women were followed up for NST in the antepartum period (18).

The results of the Non-Stress test; Variables in the external environment (such as maternal abdominal palpation, voice, and fetal sleep) may affect the procedure (4). In the literature, it has been reported that some practices such as listening to music while applying the Non-Stress test, relaxation exercises and relaxation training increase the Reactive (Negative) Non-Stress Test result expected in fetal well-being, increase the average number of accelerations, and cause a significant decrease in the level of anxiety in pregnant women (1,3,6,12,13,19,21-25). It was reported that the mean number of accelerations was 8.9±3.9 in pregnant women who were listened to music during NST application, and 4.3±3.2 in pregnant women who were not listened to. Again, in this study, NST results were reported as reactive in 98.0% of pregnant women who were listened to music and 66% of those who were not listened to (6). Similarly, while Küçükkelepçe and Timur Taşhan's (2018) average number of accelerations while listening to music was 2.14 ± 1.12, the average number of accelerations in the control group was 1.29 ± 1.09. reported (19). In addition, in the study of In the study of one in which they examined the effect of relaxation training on the reactivity of NST, they reported that the rate of reactive NST in relaxation training was 53.2%, while the rate of non-reactive NST was 46.8% (1). Based on these studies in the literature, it is seen that these practices within the scope of midwifery care practices have an effect on the NST results. In recent years, virtual reality glasses application as one of these applications has taken its place in the literature. Although virtual reality glasses technology is a device, it has been widely used in the medical field in hospitals. When the literature is examined, it is seen that virtual reality glasses reduce the level of anxiety and reduce the perception of fatigue level (20, 7, 10, 11). In the literature, in a meta-analysis study on the effectiveness of VR glasses on pain and anxiety in pediatric patients undergoing medical procedures, it was reported to be effective in reducing anxiety (SMD = 1.32; 95% CI, 0.21-2.44; P = .020) (29). In another meta-analysis, it is seen that virtual reality glasses are effective in reducing pre-operative anxiety (30) Again,one in the study of It has been reported that they have pre-anxiety anxiety and that virtual reaIn the study of onelity glasses can be a potential tool to provide low perception of fatigue levels (20).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45,
* Healthy pregnant women,
* No cardiovascular disease diagnosed in the fetus,
* Having completed the 32nd gestational week,
* Having eaten at least two hours before the NST procedure,
* Not smoking or consuming alcohol at least two hours before the NST procedure,
* Pregnant women who have no communication and visual impairments were included in the study.

Exclusion Criteria:

* • Pregnant women with fetal distress and for whom emergency intervention is considered by the physician,

  * Pregnant women with impaired NST and needing intervention at that time,
  * Pregnant women with uterine contraction as a result of NST were excluded from the study.

Ages: 32 Weeks to 40 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — pregnant
Enrollment: 87 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
When virtual reality glasses are applied during the Non-Stress test application; (1) increase fetal heart rate and fatal heart rate? | through study completion, wenty minutes
  occurring at least 2 times within a maximum of 20 minutes, at least 15 beats/min more than basal level and lasting for 15 seconds
When virtual reality glasses are applied during the Non-Stress test application; (2) increases maternal satisfaction? | through study completion, twenty minutes
  The scale is a 5-point Likert-type scale consisting of 19 items including nursing care. All items of the Newcastle Nursing Care Satisfaction Scale are positive. In the scoring used to determine the degree of satisfaction, there are statements such as "Not at all Satisfied=1 point, Slightly Satisfied=2 points, Fairly Satisfied=3 points, Very Satisfied=4 points, Extremely Satisfied=5 points". The scores given to the questions of all items marked on the score evaluation scale are added together. The maximum score obtained from the scale is 95, and the minimum score is 19. Evaluation is made by converting the total score obtained from the scale to 100. The increase in the total score obtained from the scale indicates that the patients' satisfaction with nursing is high.
When virtual reality glasses are applied during the Non-Stress test application; Does it reduce the level of maternal anxiety? | through study completion, twenty minutes
  Scoring in the State Anxiety Scale varies between 20-80 points. A score of less than 36 is considered no anxiety, a score of 37-42 is considered mild anxiety, and a score of 42 and above is considered high anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- TurkishMoHKahramanmarasPH, Kahramanmaraş, Onikişubat, Turkey (Türkiye)